CLINICAL TRIAL: NCT06308445
Title: Safety Study for the Use of Rapamycin in Children With Familial Adenomatous Polyposis.
Acronym: RAPA-4-PAF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/23/0388
Record Dates: First submitted 2024-02-22; First posted 2024-03-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Safety use; rapamycin; prophylaxis; teenager
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rapamycin (Experimental)
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — This is a 2-dose rapamycin safety study, with a target through level of 3 to <5 ng/ml for the first 3 months and 5-8 ng/ml for the next 3 months for each of the included patients. To avoid the possible cumulative effect, the two treatment phases will be separated by a 3-weeks wash-out period.

SUMMARY:
The hypothesize of this research is that rapamycin is effective and well-tolerated in teenagers with familial adenomatous polyposis (FAP). Rapamycin could be effective in blocking the formation of adenomas and/or their evolution by decreasing their size and number. Researchers aim to assess the safety profile of rapamycin in FAP adolescents using a 2 low dose regimen.

DETAILED DESCRIPTION:
FAP is a rare genetic disease linked to mutations of APC gene. Adenomatous polyps appear around the age of 10 and will evolve into colic adenocarcinoma. To date, there is no effective treatment; 100% of patients will develop colorectal cancer before 40 years. This risk is addressed by regular colonoscopy monitoring, in order to propose a timely prophylactic colectomy.

Rapamycin (sirolimus) is a drug that targets the mTOR (mammalian target of rapamycin) protein involved in the PI3K-Akt signalling pathway downstream of PI3K. There are interactions between the PI3K-Akt pathway and the Wnt/APC/-catenin pathway that is hyperactivated in FAP. Rapamycin was used out of indication with efficacy and good tolerance in 2 adolescents whose parents had refused colectomy. Researchers recently demonstrated its effectiveness in a child with very severe juvenile polyposis. Data are also available in animals, but no proof-of-concept studies have been conducted in humans.

In France, Rapamycin use is allowed in adults with kidney transplantation and pulmonary lymphangioleiomyomatosis. However, it is used on children over the market. According to the literature and the field experience, the hypothesize is that a through level of 3-8 ng/ml should be effective in children with FAP, with a lower rate of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12 to 17 at time of inclusion.
* Patients with colonoscopy for diagnosis or follow-up of FAP.
* ≥ 5 polyps (> 2 mm) at initial colonoscopy (V1).
* Free and informed consent, signed by both holders of parental authority/legal representative, with the accord of the minor patient.
* Affiliated with a social security scheme.
* Patients of childbearing potential must agree to the use of a method of contraception during the study.

Exclusion Criteria:

* Inability to understand the nature and goals of the study and/or communication difficulties observed by the investigator.
* Contraindication to performing a colonoscopy.
* < 5 polyps (>2 mm) registered during initial colonoscopy (V1).
* Advanced disease with high-grade dysplasia adenoma or even adenocarcinoma in situ that should required colectomy
* Signs of primary tuberculosis infection or respiratory infection
* Any other medical or psychological condition deemed incompatible with the proper conduct of the study according to the investigator.
* Contraindications to rapamycin use
* Participation in other biomedical research
* Deprivation of liberty of the legal guardians by judicial or administrative decision.
* Pregnancy, breastfeeding

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the safety profile of two doses of rapamycin in adolescents with Familial Adenomatous Polyposis. | For the entire duration of taking the experimental drug (rapamycin) and up to one month after stopping.
  Monitoring of adverse events (EvI) and serious adverse events (SvIG). Particular attention will be paid to known adverse events attributable to rapamycin according to the summary of product characteristics (SmPC).

SECONDARY OUTCOMES:
Evaluation of the effect of rapamycin on the number of polyps, on the entire colon and by segments (rectum, left colon, transverse colon and right colon) in adolescents suffering from Familial Adenomatous Polyposis | Visit 1 inclusion and 6 month after
  Analysis of the colonoscopies individually, blinded to the identity of the patient and the temporality of the colonoscopy in relation to the treatment, allowing a descriptive analysis of the number of polyps per segment (rectum, left colon, transverse colon, right colon).
Evaluation of the effect of rapamycin on the size of polyps, on the entire colon and by segments (rectum, left colon, transverse colon and right colon) in adolescents suffering from Familial Adenomatous Polyposis. | Visit 1 inclusion and 6 month after
  Analysis of the colonoscopies individually, blinded to the identity of the patient and the temporality of the colonoscopy in relation to the treatment, allowing a descriptive analysis of the size of polyps per segment (rectum, left colon, transverse colon, right colon).
Evaluation of the effect of rapamycin on the size of the largest polyp in each segment (rectum, left colon, transverse colon and right colon) in adolescents with Familial Adenomatous Polyposis | After 6 months of treatment with rapamycin
  Colonoscopies will be analyzed in a paired manner for each patient (before treatment / after treatment) in order to be able to make a more specific judgment of the evolution of the polyps.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mas, Pr, Study Chair — University Hospital, Toulouse
Locations (4):
- France (4):
  - CHU Bordeaux Hôpital Pellegrin, Bordeaux
  - CHU Montpellier Hôpital Arnaud de Villeneuve, Montpellier
  - APHP Hôpital Robert Debré, Paris
  - CHU Toulouse Hôpital des Enfants, Toulouse

IPD SHARING:
Plan to Share IPD: No